CLINICAL TRIAL: NCT06158932
Title: A Single Group Study to Evaluate the Effects of a Myo-Inositol and D-Chiro Inositol Supplement on Symptoms Associated With Polycystic Ovary Syndrome and Hormone Imbalance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optify (Other)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20366
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome; Hormone Imbalance
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myo Inositol and D-Chiro Inositol Supplement (Experimental): Participants must take 4 capsules per day, with water. The product should be taken with the last meal of the day.
  Interventions: Dietary Supplement: Optify Myo Inositol and D-Chiro Inositol Plus Folate and Vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Optify Myo Inositol and D-Chiro Inositol Plus Folate and Vitamin D supplement — This product contains Myo-Inositol, D-Chiro-Inositol, Folate and Vitamin D.

SUMMARY:
This is a virtual single group study that will last 12 weeks. 40 female participants will take 4 capsules of the Optify Myo Inositol and D-Chiro Inositol Plus Folate and Vitamin D supplement per day. Questionnaires will be completed at Baseline, Week 4, Week 8 and Week 12. Participants will also provide a waist circumference measurement at Baseline and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 - 55
* BMI less than 35
* Self-reported symptoms of PCOS like irregular periods, excessive hair growth, weight gain, oily skin, or acne
* Self-reported concerns around irregular menstrual cycles and ovulation, mood swings, stress, irritability, and low energy
* Self-reported concerns with hormonal skin issues
* Has access to a tape measure for waist measurement
* Generally healthy - don't live with any uncontrolled chronic disease

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone with known severe allergic reactions
* Anyone who is pregnant or breastfeeding
* Unwilling to follow the study protocol

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Changes in menstrual cycle regularity. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires with participants reporting menstrual cycle occurrence and regularity during the trial.
Changes in severity of menstrual cramps. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in hormonal skin issues. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in excessive body hair or facial hair. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.

SECONDARY OUTCOMES:
Changes in mood. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in stress. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in food cravings. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in sleep quality. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in energy. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States